CLINICAL TRIAL: NCT05730777
Title: Correlation Between Early Myocardial Injury and Intestinal Flora Changes Associated With Oncology Drug Therapy and the Preventive and Curative Effects of Probiotics
Brief Title: Correlation Between Myocardial Injury and Intestinal Flora Changes Associated With Oncology Drug Therapy and the Preventive of Probiotics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2021485
Record Dates: First submitted 2023-02-06; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Cancer Therapy-related Cardiovascular Toxicity
MeSH Terms: interventions — Probiotics; Cisplatin; Carboplatin; Paclitaxel; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium Bifidum Oral Capsule in addition to conventional treatment (Experimental): Bifidobacterium Bifidum Oral Capsule for 6 months in addition to conventional treatment
  Interventions: Drug: Bifidobacterium Bifidum Oral Capsule; Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Atlizumab
- conventional antitumor treatment (Active Comparator): Patients in the control group will receive conventional antitumor treatment only.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Paclitaxel; Drug: Atlizumab

INTERVENTIONS:
Drug: Bifidobacterium Bifidum Oral Capsule — Bifidobacterium Bifidum Oral Capsule for 6 months in addition to conventional treatment
  Other Names: Probiotics
  Arms: Bifidobacterium Bifidum Oral Capsule in addition to conventional treatment
Drug: Cisplatin — Patients in the control group will receive conventional antitumor treatment only.
  Other Names: conventional antitumor treatmen
Drug: Carboplatin — Patients in the control group will receive conventional antitumor treatment only.
  Other Names: conventional antitumor treatmen
Drug: Paclitaxel — Patients in the control group will receive conventional antitumor treatment only.
  Other Names: conventional antitumor treatmen
Drug: Atlizumab — Patients in the control group will receive conventional antitumor treatment only.
  Other Names: conventional antitumor treatmen

SUMMARY:
The purpose of this study was to explore the relationship between early myocardial injury caused by tumor drug therapy and intestinal microbial structure changes by echocardiographic two-dimensional speckle tracking technique and intestinal microflora structure detection. The investigators will also explore prevention and treatment through randomized controlled trials to initiate early intervention before clinical symptoms appear.

DETAILED DESCRIPTION:
This is a single-center randomized controlled trial in which 100 patients treated with antineoplastic agents will be enrolled. All participants will be followed for 6 months after the initiation of oncology drug therapy. Echocardiography and 2D speckle tracking will be performed and stool and blood samples will be tested before treatment initiation and at 3 and 6 months after initiation. All patients will be randomly divided into test and control groups. Patients in the test group will receive oral Bifidobacterium trivium capsules for 6 months in addition to conventional treatment, whereas patients in the control group will receive conventional antitumor treatment only.

ELIGIBILITY:
Inclusion Criteria:

* With malignant tumors
* Will receive antitumor drugs
* Could receive regular follow-up for 6 months
* Written informed consent

Exclusion Criteria:

* Satisfactory echocardiographic images could not be obtained
* Cardiomyopathy
* Coronary artery disease
* Heart failure
* Arrhythmia requiring intervention
* Moderate or severe valvular disease
* Acute myocarditis
* Refractory hypertension
* Participating in other studies of drug intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The decline rate of global longitudinal strain | 6 months
  The primary endpoint is at least a 10% decrease in the global longitudinal strain, determined using cardiac 2D STE.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Doctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No